CLINICAL TRIAL: NCT02952846
Title: Tapering of Analgosedation and Occurrence of Withdrawal Syndrome in Paediatric Intensive Care Treatment
Acronym: ASWISPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Gunnar Bentsen, Consultant, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016_ASWISPIC
Record Dates: First submitted 2016-08-30; First posted 2016-11-02 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Drug Withdrawal Symptoms; Critical Care; Child
MeSH Terms: conditions — Substance Withdrawal Syndrome | interventions — Algorithms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Before algorithm (No Intervention): Observational
- After algorithm (Experimental): Algorithm for tapering of analgosedation
  Interventions: Other: Algorithm for tapering og analgosedation

INTERVENTIONS:
Other: Algorithm for tapering og analgosedation — Algorithm for tapering og analgosedation
  Arms: After algorithm

SUMMARY:
The study is a prospective interventional study with three main aims:

1. Describe the frequency and severity of withdrawal syndrome in a population of paediatric intensive care patients.
2. Test whether implementation of an algorithm for tapering of analgosedation changes the frequency and severity of withdrawal symptoms in the same population.
3. Investigate how the health care providers experience having to adhere to such an algorithm.

DETAILED DESCRIPTION:
Patients < 18 years of age treated in an intensive care unit for 5 days or more with infusion of opioids and/or benzodiazepines, are eligible for inclusion. Patients are included at the time tapering of these drugs is initiated. Part one of the study is observational. Drugs administered, complications, Comfort score and WAT-1 (Withdrawal Assessment Tool-1) score is recorded. Before part two of the study, an algorithm for tapering of analgosedation is implemented, and the data set is obtained as in part one.

For part three of the study, focus group interviews will be used.

ELIGIBILITY:
Inclusion Criteria:

* < 18 years
* treated in PICU
* Infusion of opioids and/or benzodiazepins for 5 days or more.

Exclusion Criteria:

* Neuromuscular disease
* Cognitive/neurological disturbance caused by a disease
* Multiple disabilities

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2016-05; Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Change in mean peak WAT-1 score | Through study completion, up to 21 days

SECONDARY OUTCOMES:
Time used tapering analgosedation | Through study completion, up to 21 days
Ventilator days | Through study completion, up to 21 days
ICU days | Through study completion, up to 21 days
Drug doses used | Through study completion, up to 21 days
Adverse events | Through study completion, up to 21 days
Comfort score | Through study completion, up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar bentsen, MD PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No